CLINICAL TRIAL: NCT00001879
Title: Collection of Blood and Stool Samples in Patients With Acute Hepatitis
Brief Title: Collections of Blood and Stool Samples in Patients With Acute Hepatitis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990060; 99-H-0060
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2000-02

CONDITIONS: Hepatitis
Keywords: Liver Disease; Novel Agents; Serum; Viruses; non-A,G Hepatitis; Seronegative Acute Hepatitis
MeSH Terms: conditions — Hepatitis; Liver Diseases; Virus Diseases

SUMMARY:
Hepatitis is an inflammation of the liver. Hepatitis can be caused by an infection with a virus, but poisonous (toxic) substances can also cause it. Researchers have identified several of the viruses responsible for hepatitis, however some patients with hepatitis show no evidence of being infected with known hepatitis viruses. Researchers call conditions like this, seronegative hepatitis. It means that a patient has hepatitis but he/she does not have evidence in their blood of a viral infection.

Seronegative hepatitis is often complicated by autoimmune disorders and associated severe disorders especially, fulminant hepatitis of childhood and post-hepatitis aplastic anemia.

Researchers have attempted to identify the cause of these conditions but have been unsuccessful. Therefore, this study was developed to collect blood and stool samples from patients with seronegative hepatitis in order to help identify the virus responsible.

DETAILED DESCRIPTION:
While several viruses have been identified as agents of liver inflammation, some proportion of cases of acute hepatitis are seronegative and show no evidence of prior infection with known hepatitis viruses A, B, C, or E. Seronegative acute hepatitis is often complicated by autoimmune phenomena or late severe consequences, especially fulminant hepatitis of childhood and post-hepatitis aplastic anemia. Efforts in the Hematology Branch to identify an infectious agent in these latter two syndromes have been unsuccessful, probably because they are immune-mediated and also accompanied by massive tissue destruction. We now propose systematic collection of blood and fecal samples from patients with seronegative acute hepatitis for purposes of virus identification research. Samples will be collected from patients in United States Army clinics; patient identifiers will be employed.

ELIGIBILITY:
Collection of blood samples.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1999-03; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Atillasoy E, Berk PD. Fulminant hepatic failure: pathophysiology, treatment, and survival. Annu Rev Med. 1995;46:181-91. doi: 10.1146/annurev.med.46.1.181. PMID 7598455
- [Background] Williams R. Classification, etiology, and considerations of outcome in acute liver failure. Semin Liver Dis. 1996 Nov;16(4):343-8. doi: 10.1055/s-2007-1007247. PMID 9027947